CLINICAL TRIAL: NCT06858046
Title: Health Impacts of Fresh Cut Street Vended Fruits: A Controlled Intervention Study
Brief Title: Health Impacts of Street Vended Fruits
Acronym: HISVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh Agricultural University (Other)
Responsible Party: Principal Investigator, Md. Ariful Islam, Prof. Dr., Bangladesh Agricultural University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AWEEC/BAU/2024(2)/15(a); AWEEC/BAU/2024(2)/15(a) (Other: Animal Welfare and Experimentation Ethics Committee, Bangladesh Agricultural University, Mymensingh 2202)
Record Dates: First submitted 2025-02-23; First posted 2025-03-05 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Diseases; Foodborne Diseases; Microbial Contamination; Street Vended Foods; S. Aureus; Escherichia Coli; Total Viable Count
Keywords: Gastrointestinal Symptoms; Food borne illness; Food safety; Food borne infection; Food poisoning; S. aureus; E. coli; Bacterial contamination; Bacterial load
MeSH Terms: conditions — Gastrointestinal Diseases; Foodborne Diseases; Staphylococcal Infections; Escherichia coli Infections

STUDY DESIGN:
Intervention Model Description: This study employs a randomized controlled intervention design with a parallel assignment model to evaluate the health impacts of consuming fresh-cut street-vended fruits, focusing on microbial contamination and gastrointestinal (GI) symptoms. A total of 300 participants will be assigned to one of seven arms: two treatment arms with 75 participants each (one with gastric acidity problems and one without), subdivided into three subgroups based on the type of fruit consumed (guava, pineapple, and watermelon). Additionally, a control group of 75 participants will not consume any fresh-cut street-vended fruits and will follow their usual dietary habits. The primary aim is to assess the microbial load (Total Viable Count, S. aureus, and E. coli) on fruits and its association with the development of GI symptoms. The study will employ statistical analysis techniques, including chi-square tests, relative risk analysis, and correlation studies, to evaluate the impact of fruit consumption on
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Control Group (No Fresh-Cut Fruit Consumption) (No Intervention): Participants in this group did not consume any street-vended fresh-cut fruits. They continued their usual dietary habits, avoiding any foods that could potentially cause irritation or foodborne illness. This group served as a baseline for comparison against the treatment groups.
- Fresh-Cut Fruit Consumers with Gastric Acidity (Guava) (Experimental): Participants with pre-existing gastric acidity conditions consumed fresh-cut guava from street vendors. Their health status was monitored for five days post-consumption, focusing on gastrointestinal (GI) symptoms and microbial contamination effects.
  Interventions: Dietary Supplement: Fresh-Cut Guava Consumption (With Gastric Acidity)
- Fresh-Cut Fruit Consumers with Gastric Acidity (Pineapple) (Experimental): Participants with pre-existing gastric acidity conditions consumed fresh-cut pineapple from street vendors. Post-consumption symptoms and microbial contamination were assessed over a five-day period.
  Interventions: Dietary Supplement: Fresh-Cut Pineapple Consumption (With Gastric Acidity)
- Fresh-Cut Fruit Consumers with Gastric Acidity (Watermelon) (Experimental): Participants with pre-existing gastric acidity conditions consumed fresh-cut watermelon from street vendors. GI symptoms and potential microbial contamination effects were monitored for five days.
  Interventions: Dietary Supplement: Fresh-Cut Watermelon Consumption (With Gastric Acidity)
- Fresh-Cut Fruit Consumers without Gastric Acidity (Guava) (Experimental): Participants without pre-existing gastric acidity conditions consumed fresh-cut guava from street vendors. Health status was tracked for five days, with a focus on microbial contamination and foodborne illness symptoms.
  Interventions: Dietary Supplement: Fresh-Cut Guava Consumption
- Fresh-Cut Fruit Consumers without Gastric Acidity (Pineapple) (Experimental): Participants without pre-existing gastric acidity conditions consumed fresh-cut pineapple from street vendors. The study monitored their health for five days to evaluate any adverse effects.
  Interventions: Dietary Supplement: Fresh-Cut Pineapple Consumption
- Fresh-Cut Fruit Consumers without Gastric Acidity (Watermelon) (Experimental): Participants without pre-existing gastric acidity conditions consumed fresh-cut watermelon from street vendors. GI symptoms and microbial contamination effects were assessed over five days.
  Interventions: Dietary Supplement: Fresh-Cut Watermelon Consumption

INTERVENTIONS:
Dietary Supplement: Fresh-Cut Guava Consumption — Participants eat a defined portion of guava.
  Arms: Fresh-Cut Fruit Consumers without Gastric Acidity (Guava)
Dietary Supplement: Fresh-Cut Pineapple Consumption — Participants consumed fresh-cut pineapple purchased from street vendors. Health outcomes, including potential microbial contamination and GI symptoms, were assessed for five days after consumption.
  Arms: Fresh-Cut Fruit Consumers without Gastric Acidity (Pineapple)
Dietary Supplement: Fresh-Cut Watermelon Consumption — Fresh-Cut Watermelon Consumption Description: Participants consumed fresh-cut watermelon obtained from street vendors. GI symptoms and microbial contamination effects were monitored for five days following consumption.
  Arms: Fresh-Cut Fruit Consumers without Gastric Acidity (Watermelon)
Dietary Supplement: Fresh-Cut Guava Consumption (With Gastric Acidity) — Same as intervention 2, but in participants with acidity
  Arms: Fresh-Cut Fruit Consumers with Gastric Acidity (Guava)
Dietary Supplement: Fresh-Cut Pineapple Consumption (With Gastric Acidity) — Same as intervention 3, but in participants with acidity.
  Arms: Fresh-Cut Fruit Consumers with Gastric Acidity (Pineapple)
Dietary Supplement: Fresh-Cut Watermelon Consumption (With Gastric Acidity) — Same as intervention 4, but in participants with acidity.
  Arms: Fresh-Cut Fruit Consumers with Gastric Acidity (Watermelon)

SUMMARY:
This study will employ a randomized controlled intervention design to evaluate the health impacts of consuming fresh-cut street-vended fruits, focusing on microbial contamination and gastrointestinal (GI) symptoms. A total of 300 participants will be recruited and divided into treatment (consuming guava, pineapple, or watermelon) and control groups (no fruit consumption). Fruit samples will be analyzed for microbial contamination, including S. aureus and E. coli, using standard microbiological and molecular techniques. Data on GI symptoms will be collected through questionnaires and analyzed using statistical methods, such as Chi-square tests, Kaplan-Meier survival analysis, and Cox proportional hazards regression. Spearman correlation will identify associations between bacterial presence and specific symptoms. Ethical approval will be obtained, and participant safety will be prioritized. Analytical tools, including IBM SPSS, RStudio, and PyCharm, will be utilized for the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-60 years.
* Residents of Mymensingh District, Bangladesh.
* Willing to consume fresh-cut street-vended fruits (guava, pineapple, or watermelon) for five consecutive days.
* Individuals with a self-reported history of gastric acidity issues (for the gastric acidity arms).
* Individuals with no history of gastric acidity (for the non-gastric acidity arms).
* Participants who have not taken antibiotics, proton pump inhibitors (PPIs), or antacids in the last two weeks.
* Willing to provide detailed information on their dietary habits and gastrointestinal symptoms through surveys/questionnaires.
* Participants who provide informed consent for participation.

Exclusion Criteria:

* Individuals under 18 years or over 60 years.
* Pregnant or lactating women.
* Those with a diagnosed gastrointestinal disorder (e.g., peptic ulcer disease, irritable bowel syndrome, Crohn's disease).
* Individuals with a history of chronic infections or immune-compromising conditions (e.g., HIV/AIDS, cancer, diabetes).
* Participants who have taken antibiotics, PPIs, or antacids within the last two weeks.
* Individuals with known allergies to guava, pineapple, or watermelon.
* Those who refuse to consume fresh-cut fruits from street vendors.
* Participants who do not provide informed consent or are unable to complete the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Prevalence of Gastrointestinal Symptoms Among Participants After Consumption of Fresh-Cut Fruits | From enrollment to the end of treatment at 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Md. Ariful Islam, PhD, Principal Investigator — Bangladesh Agricultural University, Mymensingh
Locations (1):
- Department of Microbiology and Hygiene, Bangladesh Agricultural University, Mymensingh, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided